CLINICAL TRIAL: NCT04730752
Title: Prospective Clinical Trial on Validation and Comparison of the Diagnostic and Prognostic Value of Appendicitis Inflammatory Response Score and Adult Appendicitis Score
Brief Title: Validation and Comparison of the Appendicitis Inflammatory Response Score and Adult Appendicitis Score
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Alirıza Erdoğan, Principal Investigator, Nigde Omer Halisdemir University
Other Study IDs: 2021/07
Record Dates: First submitted 2021-01-24; First posted 2021-01-29 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Acute Appendicitis; Acute Appendicitis With Rupture
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Right Low Quadrant Pain: AIR and AAS scores will be calculated for the patients with right low quadrant pain in emergency service.
  Interventions: Diagnostic Test: Appendicitis Inflammatory Response; Diagnostic Test: Adult Appendicitis Score

INTERVENTIONS:
Diagnostic Test: Appendicitis Inflammatory Response — A scoring system used to diagnose acute appendicitis. It consists of clinical findings and laboratory parameters
Diagnostic Test: Adult Appendicitis Score — A scoring system used to diagnose acute appendicitis. It consists of clinical findings and laboratory parameters

SUMMARY:
Acute appendicitis is one of the most frequent reasons of emergency laparotomy in adults. Symptoms of acute appendicitis overlap with other clinical conditions and might present as a challenge, especially in the early phases. Despite the advances and widespread use of imaging modalities, still negative laparotomies are performed with the initial diagnosis of acute appendicitis. Several scoring systems are developed by using various clinical and laboratory parameters in order to improve the diagnostic accuracy and prevent unnecessary laparotomies.

DETAILED DESCRIPTION:
In the recent guideline of World Society of Emergency Surgeons (WSES) recommendations regarding the clinical scoring systems for acute appendicitis are remarkable. It is stated that clinical scoring systems, on their own, can be used to exclude acute appendicitis and decrease negative laparotomy rates. Currently Appendicitis Inflammatory Response Score (AIR) and Adult Appendicitis Score (AAS) are the best clinically performing scoring systems. As a result, based on strong evidence the use of these two systems are recommended. Both scoring systems are developed on the basis of clinical findings and laboratory parameters.

The aim of this study is to validate both systems as well as to compare the efficiency of both systems on excluding negative laparotomies and on the determination of severity of acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to ER with right lower quadrant pain
* Patients between 18-65 years old.

Exclusion Criteria:

* Patients receiving immun-suppressive therapy
* Patients with diagnosed malignancy
* Presence of mental retardation
* Patients with previous right hemicolectomy
* Patients with previous appendectomy
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18-65 years old, presenting to ER with right lower quadrant pain.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Exclude acute appendicitis | 6 months
  The ability of the scoring systems in detecting patients without acute appendicitis presenting with right lower quadrant pain to emergency service
Predicting the severity of acute appendicitis | 6 months
  The ability of scoring systems in predicting the rate of perforation in patients with acute appendicitis

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Ömer Halisdemir University Training and Research Hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ohle R, O'Reilly F, O'Brien KK, Fahey T, Dimitrov BD. The Alvarado score for predicting acute appendicitis: a systematic review. BMC Med. 2011 Dec 28;9:139. doi: 10.1186/1741-7015-9-139. PMID 22204638
- [Background] Huckins DS, Copeland K. Diagnostic accuracy of combined WBC, ANC and CRP in adult emergency department patients suspected of acute appendicitis. Am J Emerg Med. 2021 Jun;44:401-406. doi: 10.1016/j.ajem.2020.04.086. Epub 2020 Apr 29. PMID 32482481
- [Background] Di Saverio S, Podda M, De Simone B, Ceresoli M, Augustin G, Gori A, Boermeester M, Sartelli M, Coccolini F, Tarasconi A, De' Angelis N, Weber DG, Tolonen M, Birindelli A, Biffl W, Moore EE, Kelly M, Soreide K, Kashuk J, Ten Broek R, Gomes CA, Sugrue M, Davies RJ, Damaskos D, Leppaniemi A, Kirkpatrick A, Peitzman AB, Fraga GP, Maier RV, Coimbra R, Chiarugi M, Sganga G, Pisanu A, De' Angelis GL, Tan E, Van Goor H, Pata F, Di Carlo I, Chiara O, Litvin A, Campanile FC, Sakakushev B, Tomadze G, Demetrashvili Z, Latifi R, Abu-Zidan F, Romeo O, Segovia-Lohse H, Baiocchi G, Costa D, Rizoli S, Balogh ZJ, Bendinelli C, Scalea T, Ivatury R, Velmahos G, Andersson R, Kluger Y, Ansaloni L, Catena F. Diagnosis and treatment of acute appendicitis: 2020 update of the WSES Jerusalem guidelines. World J Emerg Surg. 2020 Apr 15;15(1):27. doi: 10.1186/s13017-020-00306-3. PMID 32295644
- [Background] Andersson M, Andersson RE. The appendicitis inflammatory response score: a tool for the diagnosis of acute appendicitis that outperforms the Alvarado score. World J Surg. 2008 Aug;32(8):1843-9. doi: 10.1007/s00268-008-9649-y. PMID 18553045
- [Background] Sammalkorpi HE, Mentula P, Leppaniemi A. A new adult appendicitis score improves diagnostic accuracy of acute appendicitis--a prospective study. BMC Gastroenterol. 2014 Jun 26;14:114. doi: 10.1186/1471-230X-14-114. PMID 24970111